CLINICAL TRIAL: NCT01304121
Title: Bioactive Glass Granules as Bone Graft Substitute in Filling Material of Bone Defects
Brief Title: Bioactive Glass Granules in Filling of Bone Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Hannu T Aro, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VSSHP#2701/2007
Record Dates: First submitted 2011-02-21; First posted 2011-02-25 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Bone Tumors
Keywords: Bone tumors; Bioactive glass; Autogenous bone grafting; Allogeneic bone grafting; PET imaging
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bioactive glass (Experimental): Resorbable bioactive glass granules
  Interventions: Device: Bioactive glass (SP53P4)

INTERVENTIONS:
Device: Bioactive glass (SP53P4) — Commercial resorbable bone graft substitute (Vioxid Ltd)
  Other Names: Abmin (trademark), Vioxid Ltd

SUMMARY:
This is a randomized clinical trial that will be carried out to examine the use of bioactive glass granules (S53P4) as bone graft substitute in filling small and large bone defects as compared with autogenous and allogeneic bone grafting, respectively.

DETAILED DESCRIPTION:
This a single center randomized trial. The hypothesis of the study is that the selected synthetic bone graft (bioactive glass granules, S53P4, Vivoxid Ltd, Turku, Finland) is as good as traditional autogenous or allogeneic bone grating in filling of non-traumatic bone defects. A total of 48 patients (stratified into two groups) will be included. The underlying bone disease will include common bening and semi-malign bone tumors (such as enchondroma and giant cell tumors) as well as tumor-like conditions (such as fibrous dysplasia, fibrous cortical defect, solitary bone cysts, aneurysmatic bone cyst).

Group I (n=24) will include patients with small benign bone lesions amenable to evacuation and autogenous bone grafting as standard of care. The patients will be randomized to autogenous bone grafting or bioactive glass granule filling. The follow-up examinations up to 52 weeks will include plain X-rays at 4, 26, and 52 weeks as well as MRI ad 4 and 52 weeks.

Group II (n=24) will include patients with a large bone defect. As the selection criteria, large defects have been defined to be defects which need allogeneic bone grafting. The patients will be randomized to allogeneic bone grafting or bioactive glass granule filling. The patients will be followed up to 52 weeks. The follow-up examinations will include X-rays at 4, 26 and 52 weeks as well as PET/CT imaging and MRI at 4 weeks and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* benign bone tumor or tumor-like condition
* age 18 years or more
* signed informed consent

Exclusion Criteria:

* a history of malignancy
* a medication affecting bone metabolism
* any device (such as pace maker) as contraindication for MRI imaging
* gravidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Radiological healing | 52 weeks
  The healing of bone defects will be examined by plain X-rays and MRI

SECONDARY OUTCOMES:
Clinical recovery | 52 weeks
  The outcome of the surgical procedure (i.e. the subjective recovery of the patients) will be evaluated by means of Rand-36 scoring system
PET imaging | 52 weeks
  PET imaging will be applied to measure blood flow and metabolic activity at the surgical site

CONTACTS AND LOCATIONS:
Overall Officials: Hannu T Aro, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Background] Valimaki VV, Aro HT. Molecular basis for action of bioactive glasses as bone graft substitute. Scand J Surg. 2006;95(2):95-102. doi: 10.1177/145749690609500204. PMID 16821652
- [Background] Valimaki VV, Moritz N, Yrjans JJ, Vuorio E, Aro HT. Effect of zoledronic acid on incorporation of a bioceramic bone graft substitute. Bone. 2006 Mar;38(3):432-43. doi: 10.1016/j.bone.2005.09.016. Epub 2005 Dec 9. PMID 16338190
- [Background] Keranen P, Itala A, Koort J, Kohonen I, Dalstra M, Kommonen B, Aro HT. Bioactive glass granules as extender of autogenous bone grafting in cementless intercalary implant of the canine femur. Scand J Surg. 2007;96(3):243-51. doi: 10.1177/145749690709600310. PMID 17966751
- [Background] Zhao D, Moritz N, Vedel E, Hupa L, Aro HT. Mechanical verification of soft-tissue attachment on bioactive glasses and titanium implants. Acta Biomater. 2008 Jul;4(4):1118-22. doi: 10.1016/j.actbio.2008.02.012. Epub 2008 Mar 4. PMID 18356122
- [Background] Koort JK, Suokas E, Veiranto M, Makinen TJ, Jalava J, Tormala P, Aro HT. In vitro and in vivo testing of bioabsorbable antibiotic containing bone filler for osteomyelitis treatment. J Biomed Mater Res A. 2006 Sep 1;78(3):532-40. doi: 10.1002/jbm.a.30766. PMID 16736479
- [Background] Alm JJ, Frantzen JP, Moritz N, Lankinen P, Tukiainen M, Kellomaki M, Aro HT. In vivo testing of a biodegradable woven fabric made of bioactive glass fibers and PLGA80--a pilot study in the rabbit. J Biomed Mater Res B Appl Biomater. 2010 May;93(2):573-80. doi: 10.1002/jbm.b.31618. PMID 20229522
- [Background] Keranen P, Koort J, Itala A, Ylanen H, Dalstra M, Hupa M, Kommonen B, Aro HT. Bioceramic inlays do not improve mechanical incorporation of grit-blasted titanium stems in the proximal sheep femur. J Biomed Mater Res A. 2010 Mar 15;92(4):1578-86. doi: 10.1002/jbm.a.32494. PMID 19437438
- See also: Homepage of the clinical research unit — http://www.orthopaedics.utu.fi